CLINICAL TRIAL: NCT00072280
Title: A Pilot Phase II Study for Children With Infantile Fibrosarcoma
Brief Title: Surgery and/or Chemotherapy in Treating Children With Infantile, Congenital, or Childhood Fibrosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARST03P1; CDR0000339565 (Other: PDQ (Physician Data Query)); NCI-2012-02561 (Other: NCI); COG-ARST03P1 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Sarcoma
Keywords: childhood fibrosarcoma; nonmetastatic childhood soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Fibrosarcoma | interventions — Dactinomycin; Cyclophosphamide; Etoposide; etoposide phosphate; Ifosfamide; Vincristine; Mesna; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy plus possible surgery (Experimental): Comprised of patients with disease lesions that are initially unresectable, or resected but with resulting grossly positive margins. All patients receive vincristine sulfate, dactinomycin, and cyclophosphamide (VAC), and mercaptoethane sulfonate (MESNA). Depending on response, patients may receive ifosfamide and etoposide (IE). Filgrastim may also be given, as needed. In addition to Chemotherapy, patients may receive Conventional Surgery.
  (See Interventions section for drug dosage and administration details.)
  Interventions: Biological: dactinomycin; Drug: cyclophosphamide; Drug: etoposide; Drug: ifosfamide; Drug: vincristine sulfate; Procedure: Conventional Surgery; Biological: MESNA (mercaptoethane sulfonate); Biological: Filgrastim
- Surgery only (Experimental): Comprised of patients with initially resectable disease lesions. All patients undergo Conventional Surgery. Those with a result of clear or microscopically positive margins remain on study in this arm, for observation with no further intervention.
  Interventions: Procedure: Conventional Surgery

INTERVENTIONS:
Biological: dactinomycin — Given Slow intravenous (IV) push over 1-5 minutes, dose < 1yr 0.025 mg/kg > or = 1 yr 0.045 mg/kg (max dose 2.5 mg) on days 1,22,43 and 64
  Other Names: DACT; Actinomycin-D; Cosmegen; NSC #3053
  Arms: Chemotherapy plus possible surgery
Drug: cyclophosphamide — Given IV over 60 minutes, dose 25 mg/kg on days 1,22,43 and 64.
  Other Names: Cytoxan; NSC #26271
  Arms: Chemotherapy plus possible surgery
Drug: etoposide — Given IV over 1 hour, dose 3.3 mg/kg in normal saline (NS) 10 cc/kg (or to equal 0.4 mg/mL concentration) on days 1-5 of IE cycle.
  Other Names: ETOP; VePesid; Etopophos; VP-16; NSC #141540
  Arms: Chemotherapy plus possible surgery
Drug: ifosfamide — Given IV over 1 hour, dose 60mg/kg in D5 1/4 NS 10 cc/kg IV on days 1-5 of IE Cycle
  Other Names: Isophosphamide; Iphosphamide; Z4942; Ifex; NSC #109724
  Arms: Chemotherapy plus possible surgery
Drug: vincristine sulfate — Given IV Push over 1 minute, dose 0.05 mg/kg (max dose 2 mg) on days 1,8,15,22,29,36,43,50,57 and 64
  Other Names: Oncovin; VCR; LCR; NSC #67574
  Arms: Chemotherapy plus possible surgery
Procedure: Conventional Surgery — Applied only when lesion is resectable. Surgery is the primary means of local control in this study and reasonable attempts at achieving clear margins with an "envelope" of normal tissue should be undertaken at the initial and/or subsequent resections.
Biological: MESNA (mercaptoethane sulfonate) — Given orally. Oral daily MESNA dose is equal to at least 60% of the daily cyclophosphamide dose.
  Other Names: Sodium 2-mercaptoethane sulfonate; UCB 3983; Mesnex; NSC #113891
  Arms: Chemotherapy plus possible surgery
Biological: Filgrastim — Given IV - Only use filgrastim if chemotherapy has been delayed or modified for hematologic toxicity, or if patient experiences a significant life-threatening toxicity due to bone marrow suppression
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
  Arms: Chemotherapy plus possible surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Giving combination chemotherapy before surgery may shrink the tumor so that it can be removed. Giving combination chemotherapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well surgery and/or combination chemotherapy work in treating children with fibrosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the event-free and relapse-free survival of children with initially unresectable congenital, infantile, or childhood fibrosarcoma treated with neoadjuvant chemotherapy comprising vincristine, dactinomycin, and cyclophosphamide (VAC) before definitive local control.

Secondary

* Determine the event-free and relapse-free survival of patients initially treated with this regimen followed by observation after local control with positive microscopic margins.
* Determine the event-free and relapse-free survival of patients initially treated with this regimen followed by additional chemotherapy comprising etoposide and ifosfamide after local control with gross positive margins.
* Determine the event-free and relapse-free survival of patients treated with surgery alone.

OUTLINE: This is a pilot, multicenter study. Patients begin treatment according to lesion resectability.

Patients with resectable lesions proceed to surgery.

* Surgery: Patients undergo resection of disease lesions. Patients with clear or microscopically positive margins undergo observation only. Patients with grossly positive margins undergo re-resection if feasible. Patients with grossly positive margins after re-resection or for whom re-resection is not feasible receive chemotherapy comprising vincristine, dactinomycin, and cyclophosphamide (VAC).

Patients with unresectable lesions receive VAC chemotherapy.

* VAC chemotherapy: Patients receive vincristine intravenously (IV) on days 1, 8, and 15 and dactinomycin IV and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with disease progression after 2-4 courses of VAC chemotherapy proceed to chemotherapy comprising etoposide and ifosfamide (IE).

Patients with stable disease after 4 courses of VAC chemotherapy proceed to IE chemotherapy.

Patients with a partial response (PR) and unresectable lesions after 4 courses of VAC chemotherapy receive 2 additional courses of VAC and are then re-evaluated. Patients proceed to surgery if they continue to have a PR or achieve a complete response (CR) and lesions are now resectable.

Patients with a CR or PR and resectable lesions after 4 courses of VAC chemotherapy proceed to surgery.

Patients with stable disease, progressive disease, or a PR and unresectable lesions after 6 courses of VAC proceed to IE chemotherapy.

* IE chemotherapy: Patients receive etoposide IV over 1 hour and ifosfamide IV over 1 hour on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with a CR or PR and resectable lesions after 2-4 courses of IE chemotherapy proceed to surgery.

All patients are followed every 3 months for 6 months, every 6 months for 1 year, and then as clinically indicated.

PROJECTED ACCRUAL: A total of 60-70 patients will be accrued for this study within 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infantile, congenital, or pediatric fibrosarcoma

  * Initial biopsy or surgery performed within the past 35 days
* No evidence of distant metastases
* Available tissue for central review

PATIENT CHARACTERISTICS:

Age

* Under 2 at diagnosis

Performance status

* Zubrod Score (ECOG)

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 10.0 g/dL* NOTE: *Transfusions allowed

Hepatic

* Total bilirubin no greater than 1.5 times upper limit of normal (ULN) (patients over 4 weeks of age)

  * Patients under 4 weeks of age with an indirect hyperbilirubinemia are eligible, provided the following criteria are met:

    * At least 2 bilirubin values at separate timepoints show a decrease in measurement
    * Direct bilirubin is no greater than 20% of the total bilirubin
* Direct bilirubin no greater than 1.5 times ULN
* Alanine Aminotransferase (ALT) less than 2.5 times ULN

Renal

* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

PRIOR/CONCURRENT THERAPY:

Biologic therapy

* No concurrent sargramostim (GM-CSF)

Chemotherapy

* No prior chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior or concurrent radiotherapy except emergent radiotherapy for impending tracheal compression

Surgery

* See Disease Characteristics

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mignon Loh, MD, Study Chair — University of California, San Francisco; Anne B. Warwick, MD, MPH, Study Chair — Medical College of Wisconsin
Locations (74):
- United States (64):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - OU Cancer Institute, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Starship Children's Health, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Chemotherapy Plus Possible Surgery | Surgery Only
Started | 3 | 4
Completed | 2 | 2
Not Completed | 1 | 2
Not completed — Found ineligible | 1 | 2
Period: Follow-up
Arm/Group | Chemotherapy Plus Possible Surgery | Surgery Only
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Early termination of study | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Plus Possible Surgery | Surgery Only | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Number; unit: participants]
  Less than 6 months | 2 | 2 | 4
  6 months or more | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 5
  Canada | 1 | 0 | 1
  Australia | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Failure-free Survival (FFS) in "Chemotherapy Plus Possible Surgery" Arm
Description: Failure is defined as the occurrence of one of the following: disease progression, defined as at least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions; relapse (defined with same criteria as for disease progression) after response; or death as a first event. Data will be summarized as number of eligible patients in each of the following categories at the time of data cutoff for analyses of 5-year FFS: 1)Failed; 2)Failure-free through 5 years of follow-up; 3)Failure-free until data cutoff (if less than 5 years of follow-up); 4)Withdrew from study; 5)Lost to follow-up. NOTE: Reported data are through March 2008 (see Caveats section).
Time Frame: Study enrollment until failure, completion of follow-up, or completion of 5-year FFS analyses (up to 5 years)
Population: By protocol design, only eligible patients were considered in the evaluation for the primary outcome measure. One (1) patient was found ineligible, leaving two (2) for the analysis population.
Measure: Number; unit: participants
Arm/Group | Chemotherapy Plus Possible Surgery
Number analyzed (Participants) | 2
participants
  Failed | 1
  Failure-free through 5 years of follow-up | 0
  Failure-free at cutoff (if < 5 years follow-up) | 1
  Withdrew from study | 0
  Lost to follow-up | 0

ADVERSE EVENTS:
Description: All eligible patients were considered in the evaluation of adverse events (AEs). Three (3) patients were considered ineligible. All other patients (two on each study arm) are included in AE reporting.
Arm/Group | Chemotherapy Plus Possible Surgery | Surgery Only
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Plus Possible Surgery (N=2) | Surgery Only (N=2)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0

LIMITATIONS AND CAVEATS:
Study closed early due to slow accrual. Analysis plans were not carried out (lack of statistical precision compromised the ability to draw appropriate conclusions). Reported Primary Outcome Measure data reflects data collection through March 2008.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.